CLINICAL TRIAL: NCT01357941
Title: Prospective Study Assessing the Need for Antepartum Thromboprophylaxis in Pregnant Women With One Prior Episode of Venous Thromboembolism
Brief Title: Need for Antepartum Thromboprophylaxis in Pregnant Women With One Prior Episode of Venous Thromboembolism (VTE)
Acronym: ROCITP2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr. Shannon Bates, McMaster University Medical Centre
Other Study IDs: HHS130511
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: venous thromboembolism; thromboembolism; deep vein thrombosis; pulmonary embolism; thromboprophylaxis; thrombosis; embolism and thrombosis; cardiovascular diseases; venous thrombosis; vascular diseases; anticoagulants; hematologic agents; cardiovascular agents; enoxaparin; dalteparin; tinzaparin; pregnancy complications
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thromboembolism; Thrombosis; Embolism and Thrombosis; Cardiovascular Diseases; Vascular Diseases; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prior VTE minor transient risk factor: Pregnant women with a single prior VTE episode that was either unprovoked or associated with a minor transient risk factor - Prophylaxis with fixed-dose LMWH
- Prior VTE major transient risk factor: Pregnant women with a single prior VTE episode that was provoked by a major transient risk factor - Surveillance

SUMMARY:
Pregnant women with a prior history of venous thromboembolism (VTE) are at increased risk of recurrent VTE. Current guidelines assessing the role of prophylaxis in pregnant women with prior VTE are based primarily on expert opinion and the optimal clinical management strategy remains unclear.

This multicentre, prospective cohort study aims to test the following hypotheses:

1. Antepartum prophylaxis with fixed-dose low molecular-weight heparin (LMWH) is safe, convenient and associated with an acceptably low risk of recurrent VTE in women with a single prior episode of VTE that was either unprovoked or associated with a minor transient risk factor. (Moderate risk cohort)
2. Withholding antepartum prophylaxis is safe (recurrence risk <1%) in pregnant women with a single prior episode of VTE provoked by a major transient risk factor. (Low risk cohort)

All study patients will receive 6 weeks of postpartum prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy (positive serum or urine)
* At least 18 years of age
* History of one prior episode of VTE consisting of DVT (diagnosed by compression ultrasonography [CUS] or venography) and/or PE (diagnosed by ventilation-perfusion [V/Q] lung scintigraphy, computed tomographic pulmonary angiography [CTPA], or traditional pulmonary angiography)

Exclusion Criteria:

* Ongoing need for therapeutic anticoagulation for prevention or treatment of cardioembolic stroke
* Known high-risk thrombophilia (specifically antithrombin deficiency, protein S deficiency, protein C deficiency, homozygosity for the factor V Leiden or prothrombin G20210A mutations, antiphospholipid antibody or compound abnormalities)
* VTE within 3 months of the current pregnancy
* Clinical risk factor for initial episode of VTE, if present, not resolved (excluding pregnancy)
* Known contraindication to anticoagulation (including active, uncontrolled bleeding or major bleed within the previous 4 weeks)
* For patients with prior unprovoked VTE, contraindication to LMWH (including allergy, HIT, impaired renal function, osteoporosis)
* Geographic or social factors precluding follow-up
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive pregnant women with prior VTE diagnosed with accurate testing.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Symptomatic venous thromboembolism | antepartum period (expected average 7 months)
  Symptomatic objectively confirmed recurrent VTE, including proximal DVT, non-fatal PE, and fatal PE during antepartum period

SECONDARY OUTCOMES:
Symptomatic recurrent venous thromboembolism | antepartum period (expected average 7 months) and first 3 months postpartum
  Symptomatic recurrent VTE antepartum and within first 3 months postpartum
Symptomatic recurrent pulmonary embolism | antepartum period (expected average 7 months) and first 3 months postpartum
  Symptomatic objectively confirmed recurrent PE antepartum and within first 3 months postpartum
Thrombocytopenia or heparin-induced thrombocytopenia (HIT) | antepartum period (expected average 7 months)
  Thrombocytopenia or HIT during antepartum period
Symptomatic osteoporosis | antepartum period (expected average 7 months) and first 3 months postpartum
  Symptomatic osteoporosis antepartum and within first 3 months postpartum
Other complications | antepartum (expected average 7 months) and within first 3 months postpartum
  Other complications sufficient to stop treatment (e.g., local and systemic reactions) antepartum and within first 3 months postpartum
Pregnancy complications and outcomes | antepartum period (expected average 7 months)
  Pregnancy complications and outcomes including fetal death, pre-eclampsia, toxemia, intrauterine growth restriction, prematurity during antepartum period
Fetal anomalies | antepartum (expected average 7 months) and during first 3 months postpartum
  Fetal anomalies
Major and minor bleeding | antepartum (expected average 7 months)
  Major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Bates, MD, Principal Investigator — McMaster University Medical Centre
Locations (2):
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

REFERENCES:
- [Background] Brill-Edwards P, Ginsberg JS, Gent M, Hirsh J, Burrows R, Kearon C, Geerts W, Kovacs M, Weitz JI, Robinson KS, Whittom R, Couture G; Recurrence of Clot in This Pregnancy Study Group. Safety of withholding heparin in pregnant women with a history of venous thromboembolism. Recurrence of Clot in This Pregnancy Study Group. N Engl J Med. 2000 Nov 16;343(20):1439-44. doi: 10.1056/NEJM200011163432002. PMID 11078768